CLINICAL TRIAL: NCT00577642
Title: A Phase II Study of Bone Marker Assessment of Multiple Myeloma Patients Treated With AminoBisphosphonates
Brief Title: Bone Marker Assessment of Multiple Myeloma Patients Treated With Aminobisphosphonates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Dana-Farber Cancer Institute (Other); American Society of Clinical Oncology (Other)
Responsible Party: Principal Investigator, Noopur Raje, Director Center for Multiple Myeloma, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-144; ASCO CDA
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2017-03-10 (Actual); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Multiple Myeloma
Keywords: aminobisphosphonates
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Other): Single arm biomarker study after a single dose of zoledronic acid
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — 4mg IV over at least 15 minutes or corrected for creatinine clearance x 1
  Other Names: Zometa

SUMMARY:
The purpose of this research study is to define the time a molecule in the participants bones called NTX begins to rise after receiving treatment with bisphosphonates. NTX is measured in the urine to determine the rate of bone breakdown. Tracking this marker may help identify a more optimal dosing schedule of bisphosphonate therapy. Bisphosphonate drugs like zoledronic acid, which will be used in this study, are used to reduce pain and bone fractures in people with multiple myeloma. There is some laboratory data to suggest that they may work against myeloma. Participants will have already undergone bisphosphonate therapy and may have received zoledronic acid as treatment. Typically these agents are continued indefinitely. Due to concerns of their long-term side effects we are looking at alternate strategies for reducing the frequency of these agents.

DETAILED DESCRIPTION:
* Each participant will receive a single dose of zoledronic acid intravenously after the screening procedures.
* Participants will then return to the clinic once every month for 6 months and have the following tests and procedures performed: Medical history update; physical exam; ECOG (Eastern Cooperative Oncology Group) Performance Status; blood tests; and urine tests.
* After 6 months there will be an end of study visit, where the following procedures will take place: medical history update; bone marrow aspirate and biopsy; skeletal survey.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older
* Confirmed diagnosis of multiple myeloma(MM) by Durie and Dalmon staging criteria on IV bisphosphonate therapy with either pamidronate or zoledronic acid for 8-12 months
* MM patients in either CR (complete response) or PR (partial response) by EBMT criteria
* ECOG Performance Status of 0-2

Exclusion Criteria:

* MM patients on active anti-MM therapy (maintenance regimens allowed)
* Renal failure with serum creatinine >2mg/dL and/or creatinine clearance of <30ml/min
* Relapsed, refractory or progressive disease
* Any condition or situation that, in the opinion of the investigator, may put the subject at significant risk, confound the results of the study, or interfere significantly with the subject's participation in the study
* Hypersensitivity or any contraindication to a single dose of zoledronic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noopur Raje, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Patel CG, Yee AJ, Scullen TA, Nemani N, Santo L, Richardson PG, Laubach JP, Ghobrial IM, Schlossman RL, Munshi NC, Anderson KC, Raje NS. Biomarkers of bone remodeling in multiple myeloma patients to tailor bisphosphonate therapy. Clin Cancer Res. 2014 Aug 1;20(15):3955-61. doi: 10.1158/1078-0432.CCR-14-0434. Epub 2014 Jun 23. PMID 24958808

RESULTS

PARTICIPANT FLOW:
Groups:
- Zoledronic Acid: Single dose Zoledronic Acid (Zoledronate) 4mg IV over at least 15 minutes (or dose corrected for creatinine clearance x1) followed by Aminobisphosphonates (aBP) cessation during study period.
Period: Overall Study
Arm/Group | Zoledronic Acid
Started | 29
Completed | 28
Not Completed | 1
Not completed — Clinical Disease Progression | 1

BASELINE CHARACTERISTICS:
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 60 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 29
ISS Stage [Number; unit: participants] — International Staging System (ISS) stage
  participants
    Stage I | 11
    Stage II | 9
    Stage III | 9
Therapy [Number; unit: participants]
  Bortezomib + lenalidomide | 14
  Bortezomib + Other | 10
  Other | 5
Autologous Transplant [Count of Participants; unit: Participants]
  Yes | 13
  No | 16
Bone Lesions [Number; unit: participants]
  > 3 bone lesions | 20
  ≤ 3 bone lesions | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urinary NTX Levels Less Than or Equal to 50nmol/mmol Cr
Description: Number of participants with urinary NTX levels less than or equal to 50 nmol/mmol creatinine (Cr) for the duration of study followup, following a single dose Zoledronic Acid (Zoledronate) 4mg IV over at least 15 minutes (or dose corrected for creatinine clearance x1). Dose administration was followed by Aminobisphosphonates (aBP) treatment cessation during study period.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Zoledronic Acid: Single dose Zoledronic Acid (Zoledronate) 4mg IV over at least 15 minutes (or dose corrected for creatinine clearance x1) followed by Aminobisphosphonates (aBP) treatment cessation during study period.
Arm/Group | Zoledronic Acid
Number analyzed (Participants) | 29
Participants
  NTX level ≤ 50 nmol/mmol Cr | 28
  NTX level > 50 nmol/mmol Cr | 1
Statistical Analysis 1: Comparison: Zoledronic Acid; Paired t-tests were used to compare differences of NTX cytokine levels at study entry versus end-of-study; Test type: Other — single group; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Single Arm Study: This was a nonintervention biomarker study after a single dose of Zoledronic acid.
Arm/Group | Single Arm Study
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Only 6 month biomarker data--but sufficient to change dosing regimen

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No